CLINICAL TRIAL: NCT03734016
Title: A Phase 3, Randomized Study of Zanubrutinib (BGB-3111) Compared With Ibrutinib in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: A Study of Zanubrutinib (BGB-3111) Versus Ibrutinib in Participants With Relapsed/Refractory Chronic Lymphocytic Leukemia
Acronym: ALPINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-305; 2018-001366-42 (EudraCT Number); CTR20190098 (Registry Identifier: ChinaDrugTrials.org)
Record Dates: First submitted 2018-11-02; First posted 2018-11-07 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; CLL; SLL; relapsed; refractory
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — zanubrutinib; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zanubrutinib (Experimental): Participants received 160 mg zanubrutinib orally twice daily until disease progression, intolerable toxicity, initiation of alternative anticancer therapy, investigator/Sponsor decision, need for prohibited medication, study withdrawal, or pregnancy.
  Interventions: Drug: Zanubrutinib
- Ibrutinib (Active Comparator): Participants received Ibrutinib 420 mg orally once daily until disease progression, intolerable toxicity, initiation of alternative anticancer therapy, investigator/Sponsor decision, need for prohibited medication, study withdrawal, or pregnancy.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Zanubrutinib — 160 mg orally twice daily
  Other Names: BGB-3111; Brukinsa
  Arms: Zanubrutinib
Drug: Ibrutinib — Ibrutinib 420 mg orally once daily
  Other Names: Imbruvica
  Arms: Ibrutinib

SUMMARY:
This study is designed to compare the overall response rate of zanubrutinib versus ibrutinib in participants with relapsed/refractory chronic lymphocytic leukemia or small lymphocytic lymphoma.

DETAILED DESCRIPTION:
This is a global, Phase 3, randomized study of zanubrutinib versus ibrutinib in 652 participants with relapsed/refractory chronic lymphocytic leukemia or small lymphocytic lymphoma.

The primary efficacy endpoint is overall response rate determined by investigator assessment. Participants were randomized in a 1:1 manner to either zanubrutinib or ibrutinib. Treatment with zanubrutinib and ibrutinib was open label.

ELIGIBILITY:
Key Inclusion Criteria

1. Confirmed diagnosis of CLL or SLL that meets the 2008 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria
2. CLL/SLL requiring treatment per 2008 IWCLL criteria
3. Relapsed or refractory to at least 1 prior systemic therapy for CLL/SLL
4. Measurable disease by computerized tomography (CT)/magnetic resonance imaging (MRI)
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
6. Life expectancy ≥ 6 months
7. Adequate bone marrow function
8. Adequate renal and hepatic function

Key Exclusion Criteria

1. Known prolymphocytic leukemia or history of, or currently suspected, Richter's transformation
2. Clinically significant cardiovascular disease.
3. Prior malignancy within the past 3 years, except for curatively treated basal or squamous cell skin cancer, non-muscle-invasive bladder cancer, carcinoma in situ of the cervix or breast
4. History of severe bleeding disorder or history of spontaneous bleeding requiring blood transfusion or other medical intervention
5. History of stroke or intracranial hemorrhage within 180 days before first dose of study drug
6. Severe or debilitating pulmonary disease
7. Active fungal, bacterial, and/or viral infection requiring systemic therapy
8. Known central nervous system involvement by leukemia or lymphoma
9. Known infection with HIV or active viral hepatitis B or C infection
10. Moderate or severe hepatic impairment, ie, Child-Pugh class B or C
11. Major surgery within 4 weeks of the first dose of study drug
12. Prior treatment with a (Burton's Kinase) BTK inhibitor
13. Toxicity from prior anticancer therapy that has not recovered to ≤ Grade 1
14. Pregnant or lactating women
15. Vaccination with a live vaccine within 35 days prior to the first dose of study drug
16. Hypersensitivity to zanubrutinib, ibrutinib, or any of the other ingredients in either drug
17. Concurrent participation in another therapeutic clinical trial

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (115):
- United States (30):
  - Carti Cancer Center, Little Rock, Arkansas
  - David Geffen School of Medicine At UCLA, Los Angeles, California
  - Rocky Mountain Cancer Centers Boulder, Boulder, Colorado
  - Scri Florida Cancer Specialists South, Fort Myers, Florida
  - Scri Florida Cancer Specialists North, St. Petersburg, Florida
  - Augusta University, Augusta, Georgia
  - Norton Cancer Institute Pavilion, Louisville, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Forrest General Hospital Cancer Center, Hattiesburg, Mississippi
  - Scri Hca Midwest Health, Kansas City, Missouri
  - Nebraska Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Atlantic Health System, Morristown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Columbia University Medical Center, New York, New York
  - Clinical Research Alliance, Inc, Westbury, New York
  - Duke University Hospital, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Willamette Valley Cancer Center, Springfield, Oregon
  - Scri Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Texas Oncology Fort Worth Cancer Center, Fort Worth, Texas
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Texas Oncology San Antonio Medical Center Usor, San Antonio, Texas
  - Texas Oncology Tyler Longview, Tyler, Texas
  - Blue Ridge Cancer Care (Oncology and Hematology Associates of Southwest Virginia), Roanoke, Virginia
  - Va Puget Sound Health Care System, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical Oncology Associates, Spokane, Washington
- Australia (7):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Icon Cancer Foundation, South Brisbane, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Health, Clayton, Victoria
  - Peninsula Private Hospital, Frankston, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Gasthuiszusters Antwerpen Sint Augustinus, Wilrijk, Belgium
- China (19):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Quanzhou First Affliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Provincial Wenzhou Hospital of Zhejiang, Wenzhou, Zhejiang
- Czechia (4):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Olomouc, Olomouc
  - Fakultni Nemocnice Ostrava, Ostrava
- France (6):
  - Hopital Prive Sevigne, Cesson-Sévigné
  - Centre Hospitalier Departemental de Vendee, La Roche-sur-Yon
  - Centre Hospitalier Le Mans, Le Mans
  - Chu Hopital Lyon Sud, PierreBenite
  - Centre Hospitalier Universitaire de Poitier Hopital de La Miletrie Hopital Jean Bernard, Poitiers
  - Chu Tours Hopital Bretonneau Service Pneumologie, Tours
- Germany (2):
  - Uniklinik Koln (Aor), Cologne
  - Evangelisches Krankenhaus Hamm, Hamm
- Italy (4):
  - Ospedale San Raffaele, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera Citta Della Salute E Della Scienza Di Torino, Torino
- Netherlands (2):
  - Gelre Ziekenhuizen, Apeldoorn
  - Albert Schweitzer Ziekenhuis, Nijmegen
- New Zealand (6):
  - Middlemore Clinical Trials, Auckland
  - Christchurch Hospital (Canterbury Health Laboratories), Christchurch
  - Waikato Hospital, Hamilton
  - North Shore Hospital, Takapuna
  - Tauranga Hospital, Tauranga
  - Wellington Regional Hospital (Ccdhb), Wellington
- Poland (9):
  - Interhem Opieka Szpitalna, Bialystok
  - Szpital Specjalist W Brzozowie,Podkarpacki Osrodek Onkologiczny, Brzozów
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespol Szpitali Miejskich, Chorzów
  - Copernicus Podmiot Leczniczy Sp Z Oo Wojewodzkie Centrum Onkologii, Gdansk
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Malopolskie Centrum Medyczne Sc, Krakow
  - Wojewodzki Szpital Specjalistyczny W Legnicy, Legnica
  - Wielospecjalistyczne Centrum Onkologii I Traumatologii Im M Kopernika W Lodzi, Lodz
  - Examen Sp Z Oo, Poznan
- Spain (10):
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Vall Dhebron, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Ico Girona, Girona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Virgen de La Salud, Toledo
- Sweden (2):
  - Skanes Universitetssjukhus I Lund, Lund
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Namik Kemal University, Tekirdağ, Turkey (Türkiye)
- United Kingdom (12):
  - Nhs Grampian Ppds, Aberdeen
  - Birmingham Heartlands Hospital, Birmingham
  - The Royal Bournemouth and Christchurch Hospitals Nhs Foundation, Bournemouth
  - Kent and Canterbury Hospital, Canterbury
  - St Jamess Institute of Oncology, Leeds
  - Barts Health Nhs Trust, London
  - Norfolk and Norwich University Hospitals Nhs Foundation Trust, Norwich
  - Nottingham University Hospitals Nhs Trust, Nottingham
  - Derriford Hospital, Plymouth
  - Southampton General Hospital, Southampton
  - Sunderland Royal Hospital, Sunderland
  - Genesiscare Oxford, Waterlooville

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/

REFERENCES:
- [Background] Brown JR, Eichhorst B, Hillmen P, Jurczak W, Kazmierczak M, Lamanna N, O'Brien SM, Tam CS, Qiu L, Zhou K, Simkovic M, Mayer J, Gillespie-Twardy A, Ferrajoli A, Ganly PS, Weinkove R, Grosicki S, Mital A, Robak T, Osterborg A, Yimer HA, Salmi T, Wang MD, Fu L, Li J, Wu K, Cohen A, Shadman M. Zanubrutinib or Ibrutinib in Relapsed or Refractory Chronic Lymphocytic Leukemia. N Engl J Med. 2023 Jan 26;388(4):319-332. doi: 10.1056/NEJMoa2211582. Epub 2022 Dec 13. PMID 36511784
- [Background] Hillmen P, Eichhorst B, Brown JR, Lamanna N, O'Brien SM, Tam CS, Qiu L, Kazmierczak M, Zhou K, Simkovic M, Mayer J, Gillespie-Twardy A, Shadman M, Ferrajoli A, Ganly PS, Weinkove R, Grosicki S, Mital A, Robak T, Osterborg A, Yimer HA, Salmi T, Ji M, Yecies J, Idoine A, Wu K, Huang J, Jurczak W. Zanubrutinib Versus Ibrutinib in Relapsed/Refractory Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma: Interim Analysis of a Randomized Phase III Trial. J Clin Oncol. 2023 Feb 10;41(5):1035-1045. doi: 10.1200/JCO.22.00510. Epub 2022 Nov 17. PMID 36395435
- [Result] Hillmen P, Brown JR, Eichhorst BF, Lamanna N, O'Brien SM, Qiu L, Salmi T, Hilger J, Wu K, Cohen A, Huang J, Tam CS. ALPINE: zanubrutinib versus ibrutinib in relapsed/refractory chronic lymphocytic leukemia/small lymphocytic lymphoma. Future Oncol. 2020 Apr;16(10):517-523. doi: 10.2217/fon-2019-0844. Epub 2020 Mar 24. PMID 32207333
- [Derived] Rhee JW, Lamanna N, Aldairy W, Chen L, Zhang J, Ramirez D, White WB. Hypertension in patients with chronic lymphocytic leukemia/small lymphocytic lymphoma in ALPINE: a secondary analysis. Blood Neoplasia. 2025 Aug 4;2(4):100150. doi: 10.1016/j.bneo.2025.100150. eCollection 2025 Nov. PMID 41424932
- [Derived] Brown JR, Li J, Eichhorst BF, Lamanna N, O'Brien SM, Tam CS, Qiu L, Huang R, Shi Y, Idoine A, Salmi T, Cohen AC, Shadman M. Acquired mutations in patients with relapsed/refractory CLL who progressed in the ALPINE study. Blood Adv. 2025 Apr 22;9(8):1918-1926. doi: 10.1182/bloodadvances.2024014206. PMID 39853273
- [Derived] Brown JR, Eichhorst B, Lamanna N, O'Brien SM, Tam CS, Qiu L, Jurczak W, Zhou K, Simkovic M, Mayer J, Gillespie-Twardy A, Ferrajoli A, Ganly PS, Weinkove R, Grosicki S, Mital A, Robak T, Osterborg A, Yimer HA, Wang M, Salmi T, Wang L, Li J, Wu K, Cohen A, Shadman M. Sustained benefit of zanubrutinib vs ibrutinib in patients with R/R CLL/SLL: final comparative analysis of ALPINE. Blood. 2024 Dec 26;144(26):2706-2717. doi: 10.1182/blood.2024024667. PMID 39316666
- [Derived] Zhou K, Wang T, Pan L, Xu W, Jin J, Zhang W, Hu Y, Hu J, Feng R, Li P, Liu Z, Liu P, Jing H, Gao S, Zhang H, Yu K, Wang Z, Zhu X, Sun Z, Li F, Yan D, Weng J, Fu L, Wang L, Salmi T, Wu K, Qiu L. Improved efficacy and safety of zanubrutinib versus ibrutinib in patients with relapsed/refractory chronic lymphocytic leukemia (R/R CLL) in China: a subgroup of ALPINE. Ann Hematol. 2024 Oct;103(10):4183-4191. doi: 10.1007/s00277-024-05823-8. Epub 2024 Jun 18. PMID 38888616
- [Derived] Moslehi JJ, Furman RR, Tam CS, Salem JE, Flowers CR, Cohen A, Zhang M, Zhang J, Chen L, Ma H, Brown JR. Cardiovascular events reported in patients with B-cell malignancies treated with zanubrutinib. Blood Adv. 2024 May 28;8(10):2478-2490. doi: 10.1182/bloodadvances.2023011641. PMID 38502198
- [Derived] Brown JR, Eichhorst B, Hillmen P, Jurczak W, Kazmierczak M, Lamanna N, O'Brien SM, Tam CS, Qiu L, Zhou K, Simkovic M, Mayer J, Gillespie-Twardy A, Ferrajoli A, Ganly PS, Weinkove R, Grosicki S, Mital A, Robak T, Osterborg A, Yimer HA, Salmi T, Wang MD, Fu L, Li J, Wu K, Cohen A, Shadman M. Plain language summary of zanubrutinib or ibrutinib in chronic lymphocytic leukemia that is resistant to treatment or has come back after treatment. Future Oncol. 2024 Apr;20(12):717-726. doi: 10.2217/fon-2023-0849. Epub 2023 Dec 13. PMID 38088119
- [Derived] Tam CS, Lamanna N, O'Brien SM, Qiu L, Yang K, Barnes G, Wu K, Salmi T, Brown JR. Health-related quality of life outcomes associated with zanubrutinib versus ibrutinib monotherapy in patients with relapsed/refractory chronic lymphocytic leukemia and small lymphocytic lymphoma: results from the ALPINE Trial. Curr Med Res Opin. 2023 Nov;39(11):1497-1503. doi: 10.1080/03007995.2023.2262378. Epub 2023 Oct 27. PMID 37752892

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 113 study centers in 15 countries (Australia, Belgium, China, the Czech Republic, France, Germany, Italy, the Netherlands, New Zealand, Poland, Spain, Sweden, Turkey, the United Kingdom, and the United States).
Pre-assignment Details: Participants were randomly assigned to one of two treatment groups. Randomization was stratified according to age (< 65 versus ≥ 65 years), geographic region (China vs non-China), refractory status (yes or no), and chromosome 17p deletion or TP53 mutation status (present or absent).
Groups:
- Zanubrutinib: Participants received 160 milligrams (mg) zanubrutinib orally twice daily until disease progression, intolerable toxicity, initiation of alternative anticancer therapy, investigator/Sponsor decision, need for prohibited medication, study withdrawal, or pregnancy.
Period: Overall Study
Arm/Group | Zanubrutinib | Ibrutinib
Started | 327 | 325
Received Study Drug | 324 | 324
Completed | 0 | 0
Not Completed | 327 | 325
Not completed — Sponsor Ended Study | 225 | 200
Not completed — Death | 69 | 83
Not completed — Withdrawal by Subject | 21 | 27
Not completed — Physician Decision | 1 | 12
Not completed — Lost to Follow-up | 6 | 2
Not completed — Miscellaneous | 5 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Analysis Set includes all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Zanubrutinib | Ibrutinib | Total
Number analyzed (Participants) | 327 | 325 | 652
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 126 | 125 | 251
  >=65 years | 201 | 200 | 401
Age, Continuous [Median (Full Range); unit: years] | 67.0 [35 to 90] | 68.0 [35 to 89] | 67.0 [35 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 93 | 207
  Male | 213 | 232 | 445
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 13 | 20
  Not Hispanic or Latino | 309 | 298 | 607
  Unknown or Not Reported | 11 | 14 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 47 | 44 | 91
  Black or African American | 4 | 2 | 6
  Native Hawaiian or Pacific Islander | 3 | 0 | 3
  White | 261 | 265 | 526
  Other | 2 | 2 | 4
  Multiple | 1 | 0 | 1
  Unknown/Not Reported | 9 | 12 | 21
Geographic Region [Count of Participants; unit: Participants]
  Asia | 49 | 45 | 94
  Australia/New Zealand | 28 | 30 | 58
  Europe | 198 | 191 | 389
  North America | 52 | 59 | 111
Chromosome 17p Deletion (del[17p]) and TP53 Mutation Status [Count of Participants; unit: Participants] — Deletion 17p is a chromosomal abnormality that occurs when part or all of the short arm of chromosome 17 is lost.
  The TP53 gene provides instructions for making a protein called tumor protein p53 (or p53) which acts as a tumor suppressor.
  Participants
    Del(17p) and/or TP53 mutation | 75 | 75 | 150
    Neither Del(17p) nor TP53 mutation | 251 | 250 | 501
    Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Assessed by the Investigator
Description: ORR is defined as the percentage of participants with a complete response (CR) / complete response with incomplete bone marrow recovery (CRi), nodular partial response (nPR) or partial response (PR) per investigator assessment.
  Disease response was assessed in accordance with the 2008 criteria of the International Workshop on CLL (IWCLL), with modification for treatment-related lymphocytosis in participants with CLL and in accordance with the Lugano classification in participants with SLL.
Time Frame: From randomization to the final efficacy analysis cutoff date of 08 August 2022, median time on follow-up was 29.6 months (maximum of 45.2 months).
Population: Intent To Treat (ITT) Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zanubrutinib | Ibrutinib
Number analyzed (Participants) | 327 | 325
percentage of participants | 83.5 [79.0 to 87.3] | 74.2 [69.0 to 78.8]
Statistical Analysis 1: Comparison: Zanubrutinib vs Ibrutinib; Test type: Non-Inferiority — Non-inferiority testing for ORR was performed using a stratified Wald test based on the stratified Mantel-Haenszel response ratio estimate against the non-inferiority margin of 0.8558 on the log scale; p < 0.0001, Stratified Wald test; Stratified by the randomization stratification factors (age, geographic region, refractory status, and 17p deletion and TP53 mutation status); Response ratio = 1.12, 95% CI 2-sided [1.04 to 1.22] — Response ratio is the estimated ratio of the overall response rate of the zanubrutinib arm divided by that of the ibrutinib arm
Statistical Analysis 2: Comparison: Zanubrutinib vs Ibrutinib; Test type: Superiority; p = 0.0035, Cochran-Mantel-Haenszel — Superiority testing was performed using a 2-sided stratified Cochran-Mantel-Haenszel test; [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: ORR Assessed by the Independent Review Committee (IRC)
Description: ORR is defined as the percentage of participants with a complete response (CR) / complete response with incomplete bone marrow recovery (CRi), nodular partial response (nPR) or partial response (PR) assessed by a blinded independent review committee. Overall response was assessed by the IRC for the purpose of regulatory filing with the Food and Drug Administration (FDA).
  Disease response was assessed in accordance with the 2008 criteria of the International Workshop on CLL (IWCLL), with modification for treatment-related lymphocytosis in participants with CLL and in accordance with the Lugano classification in participants with SLL.
Time Frame: as for outcome 1
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zanubrutinib | Ibrutinib
Number analyzed (Participants) | 327 | 325
percentage of participants | 86.2 [82.0 to 89.8] | 75.7 [70.7 to 80.3]
Statistical Analysis 1: Comparison: Zanubrutinib vs Ibrutinib; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Stratified Wald test; [statistical method as in outcome 1, analysis 1]; Response ratio = 1.14, 95% CI 2-sided [1.05 to 1.22] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Zanubrutinib vs Ibrutinib; Test type: Superiority — Superiority testing was performed using a 2-sided stratified Cochran-Mantel-Haenszel test; p = 0.0007, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Progression-free Survival (PFS) Assessed by the Investigator
Description: PFS is defined as the time from randomization to the date of first documentation of disease progression or death, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zanubrutinib | Ibrutinib
Number analyzed (Participants) | 327 | 325
months | NA [34.3 to NA] — Insufficient number of participants with events to estimate median and upper 95% confidence limit. | 34.2 [33.3 to NA] — Insufficient number of participants with events to estimate upper 95% confidence limit.
Statistical Analysis 1: Comparison: Zanubrutinib vs Ibrutinib; Test type: Non-Inferiority — Non-inferiority was tested with a non-inferiority margin (hazard ratio) of 1.33 with the use of a stratified Wald test based on the four randomization stratification factors; p < 0.0001, Stratified Wald test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.49 to 0.86] — Hazard ratio is the ratio of the hazard of the zanubrutinib arm divided by that of the ibrutinib arm
Statistical Analysis 2: Comparison: Zanubrutinib vs Ibrutinib; Test type: Superiority; p = 0.0024, Stratified Log-rank test; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Progression-free Survival Assessed by the Independent Review Committee
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Intent To Treat Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zanubrutinib | Ibrutinib
Number analyzed (Participants) | 327 | 325
months | NA [34.3 to NA] — Insufficient number of participants with events to estimate median and upper 95% confidence limit. | 35.0 [33.2 to 44.3]
Statistical Analysis 1: Comparison: Zanubrutinib vs Ibrutinib; Test type: Non-Inferiority — Noninferiority was tested with a noninferiority margin (hazard ratio) of 1.33 with the use of a stratified Wald test based on the four randomization stratification factors; p < 0.0001, Stratified Wald test — Stratified by the randomization stratification factors (age, geographic region, refractory status, and 17p deletion and TP53 mutation status); Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.49 to 0.86] — Hazard ratio is the ratio of the hazard of the zanubrutinib arm divided by that of the ibrutinib arm
Statistical Analysis 2: Comparison: Zanubrutinib vs Ibrutinib; Test type: Superiority; p = 0.0024, Stratified Log-rank test; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants With Atrial Fibrillation or Atrial Flutter
Description: Participants were considered as having an atrial fibrillation/flutter event if they had a treatment-emergent AE of either "atrial fibrillation" or "atrial flutter".
Time Frame: as for outcome 1
Population: The Safety Analysis Set includes all participants who received any dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zanubrutinib | Ibrutinib
Number analyzed (Participants) | 324 | 324
percentage of participants | 5.2 [3.1 to 8.3] | 13.3 [9.8 to 17.5]
Statistical Analysis 1: Comparison: Zanubrutinib vs Ibrutinib; Test type: Superiority; p = 0.0004, Chi-squared; Rate Difference = -8.0, 95% CI 2-sided [-12.4 to -3.6] — Rate difference is the zanubrutinib rate minus the ibrutinib rate

6. Secondary Outcome: Duration of Response Assessed by the Independent Review Committee
Description: DOR is defined as the time from the date that response criteria were first met to the date that disease progression was objectively documented or death, whichever occurred first, determined by independent central review. Median DOR was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Participants in the ITT Analysis Set with an objective response assessed by the IRC
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zanubrutinib | Ibrutinib
Number analyzed (Participants) | 282 | 246
months | NA [31.3 to NA] — Insufficient number of participants with events to estimate median and upper 95% confidence limit. | 33.9 [32.2 to 41.4]

7. Secondary Outcome: Duration of Response (DOR) Assessed by the Investigator
Description: DOR is defined as the time from the date that response criteria were first met to the date that disease progression was objectively documented or death, whichever occurred first, determined by investigator assessment. Median DOR was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Participants in the ITT Analysis Set with an objective response as assessed by the investigator
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zanubrutinib | Ibrutinib
Number analyzed (Participants) | 273 | 241
months | NA [31.3 to NA] — Insufficient number of participants with events to estimate median and upper 95% confidence limit. | 33.9 [33.9 to NA] — Insufficient number of participants with events to estimate upper 95% confidence limit.

8. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as the time from randomization to discontinuation of study drug due to any reason. Median time to treatment failure was estimated by the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zanubrutinib | Ibrutinib
Number analyzed (Participants) | 327 | 325
months | NA [NA to NA] — Insufficient number of participants with events to estimate median and 95% confidence interval. | NA [34.4 to NA] — Insufficient number of participants with events to estimate median and upper 95% confidence limit.
Statistical Analysis 1: Comparison: Zanubrutinib vs Ibrutinib; Test type: Other; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.41 to 0.72] — Hazard ratio is the ratio of the hazard of the zanubrutinib arm divided by that of the ibrutinib arm

9. Secondary Outcome: Rate of Partial Response With Lymphocytosis (PR-L) or Higher Assessed by the Independent Review Committee
Description: The rate of partial response with lymphocytosis or better is defined as the percentage of participants who achieved a complete response or a complete response with incomplete bone marrow recovery (CR/CRi), nodular partial response, partial response, or partial response with lymphocytosis assessed by the blinded IRC.
  Disease response was assessed per iwCLL 2008 criteria, with modification for treatment-related lymphocytosis for participants with CLL and per Lugano classification for participants with SLL.
Time Frame: as for outcome 1
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zanubrutinib | Ibrutinib
Number analyzed (Participants) | 327 | 325
percentage of participants | 91.7 [88.2 to 94.5] | 83.1 [78.5 to 87.0]

10. Secondary Outcome: Rate of Partial Response With Lymphocytosis (PR-L) or Higher Assessed by the Investigator
Description: The rate of partial response with lymphocytosis or better is defined as the percentage of participants who achieved a complete response or complete response with incomplete bone marrow recovery (CR/CRi), nodular partial response, partial response, or partial response with lymphocytosis as assessed by the investigator.
  Disease response was assessed according to the iwCLL 2008 criteria, with modification for treatment-related lymphocytosis for participants with CLL and in accordance with Lugano classification for participants with SLL.
  Partial response with lymphocytosis: blood lymphocytes decreased < 50% or increased from baseline, and otherwise meeting criteria for PR.
Time Frame: as for outcome 1
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zanubrutinib | Ibrutinib
Number analyzed (Participants) | 327 | 325
percentage of participants | 89.9 [86.1 to 93.0] | 82.5 [77.9 to 86.4]

11. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to the date of death due to any cause. Median OS was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Zanubrutinib | Ibrutinib
Number analyzed (Participants) | 327 | 325
months | NA [NA to NA] — Insufficient number of participants with events to estimate median and 95% confidence interval. | NA [NA to NA] — Insufficient number of participants with events to estimate median and 95% confidence interval.
Statistical Analysis 1: Comparison: Zanubrutinib vs Ibrutinib; Test type: Other; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.51 to 1.11] — Hazard ratio is the ratio of the hazard of the zanubrutinib arm divided by that of the ibrutinib arm

12. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status (GHS)/Quality of Life (QOL), Physical Functioning and Role Functioning Scores
Description: The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 = Not at all (best) and 4 = Very Much (worst) and 2 global health quality of life (QOL) questions answered on a 7-point scale where 1 = Very poor and 7 = Excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. Higher scores in GHS and functional scales indicate better quality of life.
Time Frame: Baseline and Weeks 24 and 48
Population: Participants in the ITT Analysis Set who completed the EORTC QLQ-C30 at Baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Zanubrutinib | Ibrutinib
Number analyzed (Participants) | 315 | 313
score on a scale
  GHS/QoL Scale at Week 24 | 8.18 [6.25 to 10.12] | 5.18 [3.20 to 7.17]
  GHS/QoL Scale at Week 48 | 7.28 [5.41 to 9.15] | 5.93 [3.97 to 7.89]
  Physical Functioning Scale at Week 24 | 6.55 [4.96 to 8.15] | 4.73 [3.08 to 6.38]
  Physical Functioning Scale at Week 48 | 5.46 [3.87 to 7.04] | 4.31 [2.65 to 5.97]
  Role Functioning Scale at Week 24 | 6.95 [4.85 to 9.06] | 6.32 [4.14 to 8.50]
  Role Functioning Scale at Week 48 | 6.81 [4.61 to 9.02] | 5.01 [2.69 to 7.33]
Statistical Analysis 1: Comparison: Zanubrutinib vs Ibrutinib; Analysis of Change from Baseline in EORTC QLQ-C30 GHS/QOL at Week 24. A linear mixed model for repeated measures (MMRM) includes the repeated measurement of the change from baseline as the dependent variable, and the treatment arm by assessment timepoint interaction, and baseline score as a covariate with an unstructured covariance matrix; Test type: Other; p = 0.0338, Mixed model for repeated measures (MMRM); Least Squares (LS) Mean Difference = 3.00, 95% CI 2-sided [0.23 to 5.77]
Statistical Analysis 2: Comparison: Zanubrutinib vs Ibrutinib; Analysis of Change from Baseline in EORTC QLQ-C30 GHS/QOL at Week 48. A linear mixed model for repeated measures (MMRM) includes the repeated measurement of the change from baseline as the dependent variable, and the treatment arm by assessment timepoint interaction, and baseline score as a covariate with an unstructured covariance matrix; Test type: Other; p = 0.3304, Mixed model for repeated measures (MMRM); LS Mean Difference = 1.34, 95% CI 2-sided [-1.37 to 4.06]
Statistical Analysis 3: Comparison: Zanubrutinib vs Ibrutinib; Analysis of Change from Baseline in EORTC QLQ-C30 Physical Functioning Scale at Week 24. A linear mixed model for repeated measures (MMRM) includes the repeated measurement of the change from baseline as the dependent variable, and the treatment arm by assessment timepoint interaction, and baseline score as a covariate with an unstructured covariance matrix; Test type: Other; p = 0.1189, Mixed model for repeated measures (MMRM); LS Mean Difference = 1.82, 95% CI 2-sided [-0.47 to 4.12]
Statistical Analysis 4: Comparison: Zanubrutinib vs Ibrutinib; Analysis of Change from Baseline in EORTC QLQ-C30 Physical Functioning Scale at Week 48. A linear mixed model for repeated measures (MMRM) includes the repeated measurement of the change from baseline as the dependent variable, and the treatment arm by assessment timepoint interaction, and baseline score as a covariate with an unstructured covariance matrix; Test type: Other; p = 0.3274, Mixed model for repeated measures (MMRM); LS Mean Difference = 1.15, 95% CI 2-sided [-1.15 to 3.44]
Statistical Analysis 5: Comparison: Zanubrutinib vs Ibrutinib; Analysis of Change from Baseline in EORTC QLQ-C30 Role Functioning Scale at Week 24. A linear mixed model for repeated measures (MMRM) includes the repeated measurement of the change from baseline as the dependent variable, and the treatment arm by assessment timepoint interaction, and baseline score as a covariate with an unstructured covariance matrix; Test type: Other; p = 0.6821, Mixed model for repeated measures (MMRM); LS Mean Difference = 0.63, 95% CI 2-sided [-2.40 to 3.66]
Statistical Analysis 6: Comparison: Zanubrutinib vs Ibrutinib; Analysis of Change from Baseline in EORTC QLQ-C30 Role Functioning Scale at Week 48. A linear mixed model for repeated measures (MMRM) includes the repeated measurement of the change from baseline as the dependent variable, and the treatment arm by assessment timepoint interaction, and baseline score as a covariate with an unstructured covariance matrix; Test type: Other; p = 0.2701, Mixed model for repeated measures (MMRM); LS Mean Difference = 1.80, 95% CI 2-sided [-1.40 to 5.00]

13. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Symptom Scales of Fatigue, Nausea and Vomiting, Pain, and Diarrhoea
Description: The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 = Not at all (best) and 4 = Very Much (worst) and 2 global health quality of life (QOL) questions answered on a 7-point scale where 1 = Very poor and 7 = Excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. Lower scores in symptom scales indicate better quality of life.
Time Frame: Baseline and Weeks 24 and 48
Population: Participants in the ITT Analysis Set who completed the EORTC QLQ-C30 at Baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Zanubrutinib | Ibrutinib
Number analyzed (Participants) | 315 | 313
score on a scale
  Fatigue Symptom Scale at Week 24 | -12.54 [-14.47 to -10.60] | -10.63 [-12.63 to -8.62]
  Fatigue Symptom Scale at Week 48 | -11.13 [-13.19 to -9.08] | -10.78 [-12.93 to -8.63]
  Nausea and Vomiting Symptom Scale at Week 24 | -1.21 [-2.03 to -0.38] | -0.92 [-1.77 to -0.07]
  Nausea and Vomiting Symptom Scale at Week 48 | -0.92 [-1.94 to 0.10] | -0.40 [-1.47 to 0.66]
  Pain Symptom Scale at Week 24 | -5.06 [-7.21 to -2.91] | -3.63 [-5.85 to -1.42]
  Pain Symptom Scale at Week 48 | -5.18 [-7.38 to -2.97] | -2.75 [-5.06 to -0.44]
  Diarrhoea Symptom Scale at Week 24 | -2.11 [-3.80 to -0.42] | -0.52 [-2.27 to 1.22]
  Diarrhoea Symptom Scale at Week 48 | -3.23 [-4.79 to -1.66] | -1.38 [-3.03 to 0.27]
Statistical Analysis 1: Comparison: Zanubrutinib vs Ibrutinib; Analysis of Change from Baseline in EORTC QLQ-C30 Fatigue Symptom Scale at Week 24. A linear mixed model for repeated measures (MMRM) includes the repeated measurement of the change from baseline as the dependent variable, and the treatment arm by assessment timepoint interaction, and baseline score as a covariate with an unstructured covariance matrix; Test type: Other; p = 0.1778, Mixed model for repeated measures (MMRM); LS Mean Difference = -1.91, 95% CI 2-sided [-4.70 to 0.87]
Statistical Analysis 2: Comparison: Zanubrutinib vs Ibrutinib; Analysis of Change from Baseline in EORTC QLQ-C30 Fatigue Symptom Scale at Week 48. A linear mixed model for repeated measures (MMRM) includes the repeated measurement of the change from baseline as the dependent variable, and the treatment arm by assessment timepoint interaction, and baseline score as a covariate with an unstructured covariance matrix; Test type: Other; p = 0.8174, Mixed model for repeated measures (MMRM); LS Mean Difference = -0.35, 95% CI 2-sided [-3.32 to 2.62]
Statistical Analysis 3: Comparison: Zanubrutinib vs Ibrutinib; Analysis of Change from Baseline in EORTC QLQ-C30 Nausea and Vomiting Symptom Scale at Week 24. A linear mixed model for repeated measures (MMRM) includes the repeated measurement of the change from baseline as the dependent variable, and the treatment arm by assessment timepoint interaction, and baseline score as a covariate with an unstructured covariance matrix; Test type: Other; p = 0.6294, Mixed model for repeated measures (MMRM); LS Mean Difference = -0.29, 95% CI 2-sided [-1.48 to 0.89]
Statistical Analysis 4: Comparison: Zanubrutinib vs Ibrutinib; Analysis of Change from Baseline in EORTC QLQ-C30 Nausea and Vomiting Symptom Scale at Week 48. A linear mixed model for repeated measures (MMRM) includes the repeated measurement of the change from baseline as the dependent variable, and the treatment arm by assessment timepoint interaction, and baseline score as a covariate with an unstructured covariance matrix; Test type: Other; p = 0.4933, Mixed model for repeated measures (MMRM); LS Mean Difference = -0.51, 95% CI 2-sided [-1.99 to 0.96]
Statistical Analysis 5: Comparison: Zanubrutinib vs Ibrutinib; Analysis of Change from Baseline in EORTC QLQ-C30 Pain Symptom Scale at Week 24. A linear mixed model for repeated measures (MMRM) includes the repeated measurement of the change from baseline as the dependent variable, and the treatment arm by assessment timepoint interaction, and baseline score as a covariate with an unstructured covariance matrix; Test type: Other; p = 0.3643, Mixed model for repeated measures (MMRM); LS Mean Difference = -1.43, 95% CI 2-sided [-4.51 to 1.66]
Statistical Analysis 6: Comparison: Zanubrutinib vs Ibrutinib; Analysis of Change from Baseline in EORTC QLQ-C30 Pain Symptom Scale at Week 48. A linear mixed model for repeated measures (MMRM) includes the repeated measurement of the change from baseline as the dependent variable, and the treatment arm by assessment timepoint interaction, and baseline score as a covariate with an unstructured covariance matrix; Test type: Other; p = 0.1363, Mixed model for repeated measures (MMRM); LS Mean Difference = -2.43, 95% CI 2-sided [-5.62 to 0.77]
Statistical Analysis 7: Comparison: Zanubrutinib vs Ibrutinib; Analysis of Change from Baseline in EORTC QLQ-C30 Diarrhoea Symptom Scale at Week 24. A linear mixed model for repeated measures (MMRM) includes the repeated measurement of the change from baseline as the dependent variable, and the treatment arm by assessment timepoint interaction, and baseline score as a covariate with an unstructured covariance matrix; Test type: Other; p = 0.2001, Mixed model for repeated measures (MMRM); LS Mean Difference = -1.59, 95% CI 2-sided [-4.01 to 0.84]
Statistical Analysis 8: Comparison: Zanubrutinib vs Ibrutinib; Analysis of Change from Baseline in EORTC QLQ-C30 Diarrhoea Symptom Scale at Week 48. A linear mixed model for repeated measures (MMRM) includes the repeated measurement of the change from baseline as the dependent variable, and the treatment arm by assessment timepoint interaction, and baseline score as a covariate with an unstructured covariance matrix; Test type: Other; p = 0.1121, Mixed model for repeated measures (MMRM); LS Mean Difference = -1.85, 95% CI 2-sided [-4.12 to 0.43]

14. Secondary Outcome: Change From Baseline in European Quality of Life 5-dimensions 5-levels Health Questionnaire (EQ-5D-5L) Visual Analog Scale (VAS)
Description: The EQ-5D-5L VAS measures a participant's self-rated health on a scale from 0 to 100, where 100 is 'the best health you can imagine' and 0 is 'the worst health you can imagine.' A higher score indicates better health outcomes.
Time Frame: Baseline and Weeks 24 and 48
Population: Participants in the ITT Analysis Set who completed the EQ-5D-5L VAS at Baseline; participants with available data at baseline and the relevant post-baseline visit are included in the analysis at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zanubrutinib | Ibrutinib
Number analyzed (Participants) | 315 | 315
score on a scale
  Week 24: number analyzed (Participants) | 278 | 260
  Week 24 | 7.92 (18.245) | 3.44 (16.972)
  Week 48: number analyzed (Participants) | 276 | 254
  Week 48 | 7.75 (18.806) | 3.92 (16.778)

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: An adverse event is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study drug, whether considered related to study drug or not.
  A serious adverse event (SAE) is any untoward medical occurrence that, at any dose:
  * Resulted in death
  * Was life-threatening
  * Required hospitalization or prolongation of existing hospitalization
  * Resulted in disability/incapacity
  * Resulted in a congenital anomaly/birth defect
  * Was considered a significant medical AE by the investigator based on medical judgment
Time Frame: From first dose of study drug up to 30 days after last dose, up to the end of study data cutoff (28 February 2024); median (range) time on treatment was 41.2 (0.4-59.1) months in the zanubrutinib arm and 37.8 (0.1-60.4) months in the ibrutinib arm.
Population: The Safety Analysis Set includes all participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Zanubrutinib | Ibrutinib
Number analyzed (Participants) | 324 | 324
Participants
  Any TEAE | 322 | 323
  Serious adverse events | 172 | 196

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected through the end of study, maximum time on study was 60.5 months. Adverse events were collected up to 30 days after last dose, up to the end of study data cutoff (28 February 2024); median (range) time on treatment was 41.2 (0.4-59.1) months in the zanubrutinib arm and 37.8 (0.1-60.4) months in the ibrutinib arm.
Description: All-cause mortality is reported for all randomized participants. Adverse events are all reported for all participants who received any dose of study drug.
Arm/Group | Zanubrutinib | Ibrutinib
All-Cause Mortality (participants affected / at risk) | 69/327 | 83/325
Serious Adverse Events (participants affected / at risk) | 172/324 | 196/324
Other Adverse Events (participants affected / at risk) | 310/324 | 314/324
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zanubrutinib (N=324) | Ibrutinib (N=324)
Anaemia (Blood and lymphatic system disorders) | 5 (8) | 4 (4)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hypoglobulinaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Splenic haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (3)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 11 (11)
Atrial flutter (Cardiac disorders) | 1 (1) | 2 (3)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 1 (2)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Dilated cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 3 (4)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (5) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Bronchogenic cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (4)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Large intestine perforation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric panniculitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal food impaction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 4 (4) | 3 (3)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 2 (3) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 5 (6)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acinetobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Arthritis bacterial (Infections and infestations) | 1 (1) | 2 (3)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (2) | 0 (0)
COVID-19 (Infections and infestations) | 28 (35) | 20 (27)
COVID-19 pneumonia (Infections and infestations) | 33 (44) | 22 (35)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Dacryocystitis (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Encephalomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (2)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal abscess central nervous system (Infections and infestations) | 1 (1) | 0 (0)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (2) | 3 (3)
Infection (Infections and infestations) | 1 (3) | 2 (2)
Infective tenosynovitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (3)
Keratitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Keratitis fungal (Infections and infestations) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (2) | 0 (0)
Lymphadenitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 2 (2)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 24 (39) | 33 (47)
Pneumonia bacterial (Infections and infestations) | 2 (4) | 2 (2)
Pneumonia cryptococcal (Infections and infestations) | 1 (3) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (2) | 1 (2)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1) | 1 (2)
Pneumonia parainfluenzae viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 2 (3) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (3) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (6) | 3 (4)
Septic shock (Infections and infestations) | 1 (1) | 2 (3)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 2 (2) | 1 (1)
Sporotrichosis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 2 (2)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Tick-borne viral encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (8) | 10 (13)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
False positive investigation result (Investigations) | 1 (3) | 0 (0)
Platelet count decreased (Investigations) | 2 (5) | 1 (2)
White blood cell count decreased (Investigations) | 0 (0) | 1 (5)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Water intoxication (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (3)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 1 (2)
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 1 (1)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chromophobe renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mucoepidermoid carcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Neuroendocrine carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Oral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 3 (3)
Superficial spreading melanoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thymoma malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Central nervous system haemorrhage (Nervous system disorders) | 0 (0) | 1 (2)
Cerebral haemorrhage (Nervous system disorders) | 1 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (3)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 1 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (2) | 2 (2)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 3 (5)
Bladder dysplasia (Renal and urinary disorders) | 1 (3) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic organ prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulva cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary necrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zanubrutinib (N=324) | Ibrutinib (N=324)
Anaemia (Blood and lymphatic system disorders) | 53 (82) | 56 (122)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 6 (10) | 11 (13)
Neutropenia (Blood and lymphatic system disorders) | 81 (195) | 73 (162)
Thrombocytopenia (Blood and lymphatic system disorders) | 34 (90) | 35 (92)
Atrial fibrillation (Cardiac disorders) | 22 (27) | 45 (69)
Cardiac failure (Cardiac disorders) | 6 (7) | 10 (10)
Palpitations (Cardiac disorders) | 13 (19) | 14 (16)
Sinus bradycardia (Cardiac disorders) | 8 (10) | 12 (15)
Vertigo (Ear and labyrinth disorders) | 11 (11) | 6 (6)
Cataract (Eye disorders) | 18 (22) | 10 (10)
Abdominal pain (Gastrointestinal disorders) | 20 (32) | 21 (23)
Abdominal pain upper (Gastrointestinal disorders) | 14 (18) | 7 (7)
Constipation (Gastrointestinal disorders) | 24 (30) | 27 (31)
Diarrhoea (Gastrointestinal disorders) | 61 (106) | 83 (158)
Dyspepsia (Gastrointestinal disorders) | 25 (27) | 23 (32)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 15 (22) | 17 (19)
Mouth ulceration (Gastrointestinal disorders) | 5 (6) | 10 (11)
Nausea (Gastrointestinal disorders) | 29 (47) | 32 (38)
Stomatitis (Gastrointestinal disorders) | 11 (17) | 11 (18)
Toothache (Gastrointestinal disorders) | 10 (11) | 6 (9)
Vomiting (Gastrointestinal disorders) | 22 (25) | 29 (35)
Asthenia (General disorders) | 21 (30) | 13 (16)
Chest pain (General disorders) | 2 (2) | 10 (10)
Fatigue (General disorders) | 36 (43) | 49 (57)
Influenza like illness (General disorders) | 10 (28) | 7 (10)
Oedema peripheral (General disorders) | 24 (27) | 24 (31)
Peripheral swelling (General disorders) | 14 (15) | 26 (30)
Pyrexia (General disorders) | 35 (44) | 37 (50)
Hypogammaglobulinaemia (Immune system disorders) | 12 (13) | 12 (13)
Bronchitis (Infections and infestations) | 19 (22) | 26 (34)
COVID-19 (Infections and infestations) | 121 (163) | 84 (105)
COVID-19 pneumonia (Infections and infestations) | 13 (18) | 15 (20)
Cellulitis (Infections and infestations) | 12 (15) | 13 (16)
Conjunctivitis (Infections and infestations) | 7 (10) | 15 (20)
Ear infection (Infections and infestations) | 10 (12) | 4 (5)
Gastroenteritis (Infections and infestations) | 10 (10) | 6 (6)
Herpes zoster (Infections and infestations) | 11 (12) | 10 (14)
Lower respiratory tract infection (Infections and infestations) | 12 (16) | 12 (14)
Nasopharyngitis (Infections and infestations) | 20 (26) | 16 (23)
Oral herpes (Infections and infestations) | 4 (9) | 13 (17)
Paronychia (Infections and infestations) | 5 (6) | 11 (11)
Pharyngitis (Infections and infestations) | 6 (8) | 12 (18)
Pneumonia (Infections and infestations) | 33 (47) | 37 (57)
Respiratory tract infection (Infections and infestations) | 16 (20) | 7 (8)
Rhinitis (Infections and infestations) | 10 (11) | 10 (11)
Sinusitis (Infections and infestations) | 20 (26) | 16 (19)
Skin infection (Infections and infestations) | 7 (8) | 13 (16)
Upper respiratory tract infection (Infections and infestations) | 95 (155) | 64 (105)
Urinary tract infection (Infections and infestations) | 35 (68) | 31 (58)
Contusion (Injury, poisoning and procedural complications) | 49 (62) | 38 (44)
Fall (Injury, poisoning and procedural complications) | 16 (19) | 23 (27)
Skin laceration (Injury, poisoning and procedural complications) | 12 (12) | 6 (6)
Alanine aminotransferase increased (Investigations) | 12 (20) | 20 (29)
Aspartate aminotransferase increased (Investigations) | 7 (12) | 16 (23)
Blood alkaline phosphatase increased (Investigations) | 5 (8) | 10 (15)
Blood bilirubin increased (Investigations) | 8 (14) | 11 (20)
Blood creatinine increased (Investigations) | 18 (36) | 12 (21)
Blood pressure increased (Investigations) | 6 (19) | 12 (27)
Gamma-glutamyltransferase increased (Investigations) | 10 (14) | 11 (16)
Neutrophil count decreased (Investigations) | 26 (75) | 24 (69)
Platelet count decreased (Investigations) | 11 (40) | 20 (47)
Weight decreased (Investigations) | 22 (27) | 14 (20)
Decreased appetite (Metabolism and nutrition disorders) | 12 (12) | 22 (23)
Gout (Metabolism and nutrition disorders) | 4 (10) | 10 (16)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (21) | 8 (8)
Hyperuricaemia (Metabolism and nutrition disorders) | 16 (37) | 22 (37)
Hypokalaemia (Metabolism and nutrition disorders) | 24 (39) | 24 (39)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (18) | 8 (13)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 14 (15) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 54 (69) | 63 (85)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (26) | 26 (30)
Joint swelling (Musculoskeletal and connective tissue disorders) | 10 (10) | 10 (12)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 (18) | 42 (51)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (13) | 14 (14)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (5) | 12 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 (30) | 26 (30)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (18) | 17 (40)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (21) | 15 (23)
Dizziness (Nervous system disorders) | 32 (39) | 26 (28)
Headache (Nervous system disorders) | 29 (36) | 35 (46)
Paraesthesia (Nervous system disorders) | 3 (3) | 10 (12)
Syncope (Nervous system disorders) | 11 (14) | 8 (9)
Anxiety (Psychiatric disorders) | 11 (11) | 14 (22)
Insomnia (Psychiatric disorders) | 25 (27) | 26 (28)
Haematuria (Renal and urinary disorders) | 18 (23) | 13 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 46 (59) | 43 (55)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (19) | 13 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27 (46) | 24 (45)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 10 (10)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 11 (12)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 8 (16) | 12 (15)
Ecchymosis (Skin and subcutaneous tissue disorders) | 5 (5) | 11 (12)
Erythema (Skin and subcutaneous tissue disorders) | 11 (11) | 9 (10)
Petechiae (Skin and subcutaneous tissue disorders) | 32 (41) | 19 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 24 (32) | 9 (10)
Rash (Skin and subcutaneous tissue disorders) | 38 (69) | 44 (58)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (15) | 7 (10)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 8 (12) | 12 (13)
Haematoma (Vascular disorders) | 17 (23) | 14 (17)
Hypertension (Vascular disorders) | 82 (154) | 74 (155)
Hypotension (Vascular disorders) | 3 (3) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT03734016/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT03734016/SAP_002.pdf